CLINICAL TRIAL: NCT05821309
Title: Evaluation of Fecal Microbiome Changes After Antegrade Continence Enema Placement and Initiation of Bowel Flush Regimen
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Kathryn Hawa, DO, Principle Investigator, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 17083
Record Dates: First submitted 2023-04-07; First posted 2023-04-20 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Constipation
Keywords: Fecal microbiome; Malone Antegrade Continence Enema (MACE); Miralax; PEG 3350; Antegrade Continence Enema; Chronic Constipation
MeSH Terms: conditions — Constipation | interventions — polyethylene glycol 3350; Electrolytes; Golytely; Glycerol

STUDY DESIGN:
Masking Description: Only objective data in the form of fecal microbiome diversity will be obtained via 16s rRNA sequencing. Neither the participant nor the investigators will be blinded.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PEG 3350 (Experimental): Patients will receive PEG 3350 (miralax or generic equivalent) for their MACE flushes.
  Interventions: Drug: PEG 3350; Drug: Glycerin
- PEG 3350 with electrolytes (Experimental): Patients will receive PEG 3350 with electrolytes (Go-Lytely or generic equivalent) for their MACE flushes.
  Interventions: Drug: PEG-3350 with electrolytes; Drug: Glycerin

INTERVENTIONS:
Drug: PEG 3350 — The purpose of this study is to determine if a sustained change in the fecal microbiome occurs after prolonged use of an antegrade continence enema bowel flush regimen. Patients' microbiomes will be evaluated via 16s rRNA sequencing. PEG 3350 will be compared to PEG 3350 with electrolytes
  Other Names: MiraLAX or generic equivalent
  Arms: PEG 3350
Drug: PEG-3350 with electrolytes — The purpose of this study is to determine if a sustained change in the fecal microbiome occurs after prolonged use of an antegrade continence enema bowel flush regimen. Patients' microbiomes will be evaluated via 16s rRNA sequencing. PEG 3350 will be compared to PEG 3350 with electrolytes
  Other Names: GoLytely or generic equivalent
  Arms: PEG 3350 with electrolytes
Drug: Glycerin — Glycerin will be given to patients based on standard of care, at the discretion of the pediatric gastroenterology and pediatric surgery teams. Glycerin administration will not be randomized. For secondary analysis, the microbiomes of those who have and have not received glycerin will be compared.

SUMMARY:
This study will evaluate changes in the fecal microbiome in constipated pediatric patients before and after antegrade continence enema placement and initiation of antegrade enema flushes. Subjects will have their microbiome sequenced prior to placement by obtaining a fecal sample. Pre-antegrade continence enema placement results will be compared to fecal samples obtained at 0, 4, 8 months after placement of the antegrade continence enema and initiation of miralax or golytely flushes to look for changes in bacterial diversity.

DETAILED DESCRIPTION:
This is a prospective, longitudinal study of children 2 -18 years of age who undergo a clinical Malone Antegrade Continence Enema (MACE) appendicostomy or cecostomy for treatment of chronic functional constipation as defined by the Rome IV criteria. Only patients with intact motility on colonic manometry (CMS) will be included. The antegrade enema flush medication regimen will be randomized in 1:1 ratio of PEG 3350 and PEG3350 with electrolytes. The study statistician will create a blocked randomization schedule which will be uploaded into REDCap. Glycerin and stimulant laxatives will be titrated as needed by a pediatric gastroenterologist in conjunction with the pediatric general surgery team. Neither patient nor providers will be blinded to laxative randomization as objective data in the form of microbiome composition is being evaluated.

Patients will have a pre-MACE placement stool sample obtained at time of colonic motility studies and repeat stool samples collected at 1 month, 4 months and 8 months post-MACE placement and initiation of antegrade enemas. Post-MACE samples will be submitted at standard follow-up appointments. All stool samples will be self-collected by patients. Samples will be collected with the OMNIgene GUT kit which provides stabilization of DNA at room temperature for up to 60 days. Once the sample is collected by the research team, sample tubes will be stored at -80 Celsius until all samples are collected and sent for sequencing. Pre-MACE stool samples will be collected while abstaining from osmotic laxative therapy for one week. If patients do not spontaneously pass stool during the week of osmotic laxative abstention, stool will be collected from the first bowel movement after pre-CMS bowel flush with PEG 3350 with or without electrolytes has been initiated. Data regarding if stool collection occurred before or after receiving PEG 3350 with or without electrolytes for CMS bowel flush will be recorded. Patients will perform daily flushes after MACE placement and post-MACE stool samples will be collected within the first 10 minutes of flush initiation.

ELIGIBILITY:
Inclusion Criteria:

* Recalcitrant chronic functional constipation necessitating a MACE appendicostomy or cecostomy for treatment at Riley Hospital for Children
* Intact colonic motility as evidenced by CMS studies

Exclusion Criteria

* Underlying anatomic or pathologic etiology for constipation
* History of prior gastrointestinal surgery (excluding placement of G or GJ tubes)
* Underlying severe GI disease unrelated to the patient's chronic constipation
* Use within the past month of consent of probiotic supplements, prebiotic supplements or antibiotics

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 65 (Estimated)
Dates: Start 2023-06-08 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Change in Fecal Microbiome at 1 month | At baseline and 1 month post-MACE
  The purpose of this study is to determine if a sustained change in the fecal microbiome occurs after prolonged use of an antegrade continence enema bowel flush regimen. Patients' microbiomes will be evaluated via 16s rRNA sequencing
Change in Fecal Microbiome at 4 months | At baseline and 4 months post-MACE
  The purpose of this study is to determine if a sustained change in the fecal microbiome occurs after prolonged use of an antegrade continence enema bowel flush regimen. Patients' microbiomes will be evaluated via 16s rRNA sequencing
Change in Fecal Microbiome at 8 months | At baseline and 8 months post-MACE
  The purpose of this study is to determine if a sustained change in the fecal microbiome occurs after prolonged use of an antegrade continence enema bowel flush regimen. Patients' microbiomes will be evaluated via 16s rRNA sequencing

SECONDARY OUTCOMES:
Effect of Bowel Regimen Solution on Fecal Bacterial Diversity | Through study completion, approximately 8 months
  Determine whether a difference in fecal bacterial diversity determined by 16s rRNA sequencing exists between differing MACE bowel regimens of 1. Bisacodyl and PEG 3350 in electrolyte solution (GoLytely) or 2. Bisacodyl and PEG 3350 without electrolytes (Miralax).
Effect of Glycerin on Fecal Microbiome Diversity | Through study completion, approximately 8 months
  Determine whether patients receiving glycerin in addition to PEG 3350 with or without electrolytes display differences in their fecal microbiota as measured by 16s rRNA sequencing.
Effect of Redundant Sigmoid Colon on Microbiome Diversity | Through study completion, approximately 8 months
  Evaluate for differences in the fecal microbiome determined by 16s rRNA sequencing between those patients who have a redundant sigmoid colon based on barium enema results and those who do not

CONTACTS AND LOCATIONS:
Overall Officials: Kate Hawa, DO, Principal Investigator — Riley Hospital for Children
Locations (2):
- United States (2):
  - IU North Hospital, Carmel, Indiana
  - Riley Hospital for Children, Indianapolis, Indiana

IPD SHARING:
Plan to Share IPD: No